CLINICAL TRIAL: NCT01466127
Title: The Effect of Oxytocin on Fear Memory Consolidation: A Novel Intervention to Prevent PTSD
Brief Title: The Effect of Oxytocin on Fear Memory Consolidation Novel Intervention to Prevent Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth A. Hoge, MD, Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010P-002911
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Effect of oxytocin on learning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched nasal spray placebo.
  Interventions: Drug: Placebo
- Oxytocin (Experimental): Liquid intranasal oxytocin administered in a nasal spray.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Liquid metered-dose nasal spray, 30 IUs, administered once.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Matched nasal spray placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn how differences in learning under mildly-stressful circumstances may be changed by taking oxytocin. Oxytocin is a hormone made naturally in the body. The investigators will also examine the impact of any anxiety, depression, and stress related symptoms on learning processes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 65 years of age
* Score in study range on the Neuroticism-Extraversion-Openness-Five Factor Inventory (NEO-FFI)
* No current Axis I Diagnostic and Statistical Manual-IV (DSM) excluded diagnoses as determined by the Structured Clinical Interview DSM (SCID) completed within the past 4 months.
* Must be able and willing to understand study procedures and return to the clinic on two separate consecutive days for the fear-conditioning procedures.
* Subjects must be able to give informed consent and be willing and able to comply with study procedures.

Exclusion Criteria:

* Presence of a current DSM-IV Axis I diagnosis as measured by the SCID.
* A serious medical condition or other condition deemed likely to result in surgery or hospitalization, or which would make participation in the study difficult.
* Patients with a history of trauma resulting in head injury related seizures or with epilepsy (except a prior history of febrile seizures of infancy which are not exclusionary).
* Use of supplemental hormones (birth control, estrogen, testosterone, prednisone, etc) or narcotics.
* Pregnant or lactating women.
* Women of childbearing potential not using medically accepted forms of contraception.
* Current use of the excluded psychiatric medications.
* Known hypersensitivity to oxytocin
* Known hyponatremia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Hoge, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Anxiety and Traumatic Disorders, MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Oxytocin
Started | 30 | 30
Completed | 16 | 14
Not Completed | 14 | 16

BASELINE CHARACTERISTICS:
Population: Although 60 participants were enrolled, only 30 participants had usable physiological data from recording electrodes, and therefore, the only data analyzed were from these 30 participants (16 placebo and 14 oxytocin).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Oxytocin | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.9 (14.7) | 39.9 (15.8) | 35.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Differential Skin Conductance Response (SCR) During the First Two Extinction Trials
Description: Differences in skin conductance response (SCR) between the active vs. placebo conditions trials will be used to assess for the impact of oxytocin on fear acquisition and extinction. We will take a mean of the first two extinction trials to get this measure. Data was gathered in micro-Siemens and then underwent a square root transformation.
Time Frame: Day 2 of Conditioning (1 day post Day 1 of Conditioning)
Measure: Mean (Standard Deviation); unit: micro-Siemens (square rooted)
Arm/Group | Placebo | Oxytocin
Number analyzed (Participants) | 16 | 14
micro-Siemens (square rooted) | 0.15 (0.31) | 0.00 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Oxytocin; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo | Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Oxytocin (N=14)
Bloody Nose (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes